CLINICAL TRIAL: NCT02872714
Title: A Phase 2, Open-Label, Single-Agent, Multicenter Study to Evaluate the Efficacy and Safety of Pemigatinib (INCB054828) in Subjects With Metastatic or Surgically Unresectable Urothelial Carcinoma Harboring FGF/FGFR Alterations - (FIGHT-201)
Brief Title: A Study to Evaluate the Efficacy and Safety of Pemigatinib (INCB054828) in Subjects With Urothelial Carcinoma - (FIGHT-201)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 54828-201; 2016-001321-14 (EudraCT Number)
Expanded Access: NCT03906357 (No longer available)
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Results first posted 2023-03-24 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: UC (Urothelial Cancer)
Keywords: Urothelial carcinoma; fibroblast growth factor (FGF); fibroblast growth factor receptor (FGFR); FGF/FGFR alterations
MeSH Terms: conditions — Carcinoma, Transitional Cell; Acrocephalosyndactylia | interventions — pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A-ID (Intermittent Dose) Pemigatinib (Experimental): Pemigatinib in subjects with FGFR3 mutations or fusions.
  Interventions: Drug: pemigatinib
- Cohort A-CD (Continuous Dose) Pemigatinib (Experimental): Pemigatinib in subjects with FGFR3 mutations or fusions.
  Interventions: Drug: pemigatinib
- Cohort B Pemigatinib (Experimental): Pemigatinib in subjects with other FGF/FGFR alterations.
  Interventions: Drug: pemigatinib

INTERVENTIONS:
Drug: pemigatinib — Pemigatinib once a day by mouth for 2 consecutive weeks and 1 week off therapy.
  Other Names: INCB054828
  Arms: Cohort A-ID (Intermittent Dose) Pemigatinib; Cohort B Pemigatinib
Drug: pemigatinib — Pemigatinib once a day by mouth continuously.
  Other Names: INCB054828
  Arms: Cohort A-CD (Continuous Dose) Pemigatinib

SUMMARY:
The purpose of this study is to evaluate the overall response rate (ORR) of pemigatinib as a monotherapy in the treatment of metastatic or surgically unresectable urothelial carcinoma harboring FGF/FGFR alterations.

ELIGIBILITY:
Inclusion Criteria:

* 20 years and older in Japan
* Histologically documented metastatic or surgically unresectable urothelial carcinoma; may include primary site from urethra, ureters, upper tract, renal pelvis, and bladder.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Life expectancy ≥ 12 weeks.
* Radiographically measurable per RECIST v1.1.
* Documented FGF/FGFR alteration and have either 1a) failed at least 1 previous treatment for their metastatic or surgically unresectable urothelial carcinoma (ie, chemotherapy, immunotherapy) or 1b) have not received chemotherapy due to poor ECOG status or 2) have insufficient renal function.

Exclusion Criteria:

* Prior receipt of a selective FGFR inhibitor.
* Use of any potent CYP3A4 inhibitors or inducers within 14 days or 5 half-lives (whichever is shorter) before the first dose of study drug.
* Inability or unwillingness to swallow pemigatinib or significant gastrointestinal disorder(s) that could interfere with the absorption, metabolism, or excretion of pemigatinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterine Asatiani, MD, Study Director — Incyte Corporation
Locations (96):
- United States (34):
  - Arizona Oncology Associates (Wilmot), Tucson, Arizona
  - Sharp Memorial Hospital, San Diego, California
  - UCSF Helen Diller Family Comprehensive Care Center, San Francisco, California
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Calaway-Young Cancer Center at Valley View Hospital, Glenwood Springs, Colorado
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - Lahey Clinic Inc. - PARENT ACCOUNT, Burlington, Massachusetts
  - Minnesota Oncology Hematology, P.A., Woodbury, Minnesota
  - GU Research Network, Omaha, Nebraska
  - TRIO - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York Oncology Hematology, P.C., Albany, New York
  - Northwell Cancer Institute, New Hyde Park, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Compass Oncology the Northwest Cancer Specialists, Tualatin, Oregon
  - St. Luke's Hospital, Bethlehem, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology, P.A. - Austin, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons, Dallas, Texas
  - Texas Oncology, Houston, Texas
  - Texas Oncology, P.A. - Sherman, Sherman, Texas
  - Baylor Scott & White Health, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Oncology Associates - Hampton, Norfolk, Virginia
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - University of Wisconsic Hospital and Clinic, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (4):
  - UZ Antwerpen, Edegem
  - AZ Sint-Lucas - Campus Sint-Lucas, Ghent
  - AZ Groeninge Campus Loofstraat, Kortrijk
  - AZ Delta, Roeselare
- Rigshospitalet, Copenhagen, Denmark
- France (10):
  - CHU Besançon - Hôpital Jean Minjoz, Besançon, Doubs
  - Groupe Hospitalier Saint André - Hôpital Saint André, Bordeaux, Gironde
  - Institut Claudius Regaud-Oncopole, Toulouse, Haute Garonne
  - ICO - Site René Gauducheau, Saint-Herblain, Loire Atlantique
  - ICO - Site Paul Papin, Angers, Maine Et Loire
  - Hopital Saint Louis, Paris, Paris
  - Centre Leon Berard, Lyon, Rhone
  - CHU Strasbourg - Nouvel Hôpital Civil, Strasbourg, Rhone
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (9):
  - Charite Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - Klinikum Dresden Standort Dresden-Friedrichstadt, Dresden
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Universitaetsklinikum Muenster, Münster
  - Studienpraxis Urologie Drs. Feyerabend, Nürtingen
  - Universitaetsklinikum Tuebingen, Tübingen
- Israel (5):
  - Soroka University Medical Center, Beersheba
  - Assaf Harofeh Medical Center, Be’er Ya‘aqov
  - Meir Medical Center, Kfar Saba
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (9):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Fondazione Del Piemonte Per L'Oncologia IRCC Candiolo, Candiolo
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera Di Rilievo Nazionale A. Cardarellio, Napoli
  - Ospedale degli Infermi, Rimini
  - University Campus Bio-Medico di Roma, Rome
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
  - San Camillo-Forlanini Hospital, Siena
- Japan (10):
  - Kyushu University Hospital, Fukuoka
  - Saitama Medical University International Medical Center, Hidaka-shi
  - Hirosaki University Hospital, Hirosaki-shi
  - Teikyo University Hospital, Itabashi-ku
  - Nihon University Itabashi Hospital, Itabashi-ku
  - Nara Medical University Hospital, Kashihara-shi
  - Osaka International Cancer Institute, Osaka
  - Saitama Cancer Center, Saitama
  - Osaka University Hospital, Suita-shi
  - Jichi Medical University Hospital, Tochigi
- Netherlands (4):
  - VU Medisch Centrum, Amsterdam
  - Zorgsaam Ziekenhuis, Terneuzen
  - HagaZiekenhuis Van Den Haag, The Hague
  - Viecuri Medisch Centrum, Venlo
- Spain (4):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron, Barcelona
  - ICO Girona - Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Centro Integral Oncologico Clara Campal, Madrid
- United Kingdom (6):
  - University College London Hospitals, London, Greater London
  - Guy's Hospital, London, Greater London
  - Charing Cross Hospital, London, Greater London
  - Nottingham University Hospitals City Campus, Nottingham, Nottinghamshire
  - Beatson West of Scotland Cancer Centre, Glasgow, Strathclyde
  - Queen Elizabeth Hospital, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- [Derived] Zhang C, Huang MN, Shan JQ, Hu ZJ, Li ZW, Liu JY. Pemigatinib, a selective FGFR inhibitor overcomes ABCB1-mediated multidrug resistance in cancer cells. Biochem Biophys Res Commun. 2024 Jan 8;691:149314. doi: 10.1016/j.bbrc.2023.149314. Epub 2023 Nov 24. PMID 38039831
- [Derived] Necchi A, Pouessel D, Leibowitz R, Gupta S, Flechon A, Garcia-Donas J, Bilen MA, Debruyne PR, Milowsky MI, Friedlander T, Maio M, Gilmartin A, Li X, Veronese ML, Loriot Y. Pemigatinib for metastatic or surgically unresectable urothelial carcinoma with FGF/FGFR genomic alterations: final results from FIGHT-201. Ann Oncol. 2024 Feb;35(2):200-210. doi: 10.1016/j.annonc.2023.10.794. Epub 2023 Nov 11. PMID 37956738

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted at a total of 73 study centers in 11 countries (United States, France, Italy, Spain, Israel, Belgium, United Kingdom, Germany, Japan, Denmark, and the Netherlands).
Groups:
- Cohort A-ID: FGFR3 Mutations or Fusions: Participants with fibroblast growth factor (FGF) receptor 3 (FGFR3) mutations or fusions self-administered oral pemigatinib at a starting dose of 13.5 milligrams (mg) once daily (QD) on an intermittent dose (ID) (2-weeks-on/1-week-off therapy) schedule in 21-day cycles. Participants who did not reach the target serum phosphate level of > 5.5 mg/deciliter (dL) could have increased the daily dose to 18 mg, provided they had no ongoing Grade 2 or higher treatment-related treatment-emergent adverse events (TEAEs), and they had been compliant with taking the study drug.
- Cohort B-ID: All Other FGF/FGFR Alterations: Participants with all other FGF/FGFR alterations self-administered oral pemigatinib at a starting dose of 13.5 mg QD on an ID (2-weeks-on/1-week-off therapy) schedule in 21-day cycles. Participants who did not reach the target serum phosphate level of > 5.5 mg/dL could have increased the daily dose to 18 mg, provided they had no ongoing Grade 2 or higher treatment-related TEAEs, and they had been compliant with taking the study drug.
- Other-ID: Participants with no FGF/FGFR alterations or with an undetermined FGF/FGFR status self-administered oral pemigatinib at a starting dose of 13.5 mg QD on an ID (2-weeks-on/1-week-off therapy) schedule in 21-day cycles. Participants who did not reach the target serum phosphate level of > 5.5 mg/dL could have increased the daily dose to 18 mg, provided they had no ongoing Grade 2 or higher treatment-related TEAEs, and they had been compliant with taking the study drug.
- Cohort A-CD: FGFR3 Mutations or Fusions: Participants with FGFR3 mutations or fusions self-administered oral pemigatinib at a starting dose of 13.5 mg QD on a continuous dose (CD) (no planned dose hold) schedule in 21-day cycles. Participants who did not reach the target serum phosphate level of > 5.5 mg/dL could have increased the daily dose to 18 mg, provided they had no ongoing Grade 2 or higher treatment-related TEAEs, and they had been compliant with taking the study drug.
- Other-CD: Participants with no FGF/FGFR alterations or with an undetermined FGF/FGFR status self-administered oral pemigatinib at a starting dose of 13.5 mg QD on a continuous dose (CD) (no planned dose hold) schedule in 21-day cycles. Participants who did not reach the target serum phosphate level of > 5.5 mg/dL could have increased the daily dose to 18 mg, provided they had no ongoing Grade 2 or higher treatment-related TEAEs, and they had been compliant with taking the study drug.
Period: Overall Study
Arm/Group | Cohort A-ID: FGFR3 Mutations or Fusions | Cohort B-ID: All Other FGF/FGFR Alterations | Other-ID | Cohort A-CD: FGFR3 Mutations or Fusions | Other-CD
Started | 103 | 44 | 9 | 101 | 3
Completed | 10 | 2 | 1 | 13 | 1
Not Completed | 93 | 42 | 8 | 88 | 2
Not completed — Progressive Disease | 1 | 2 | 0 | 0 | 0
Not completed — Death | 87 | 36 | 8 | 81 | 2
Not completed — Lost to Follow-up | 2 | 1 | 0 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 2 | 0
Not completed — Captured as Other | 2 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A-ID: FGFR3 Mutations or Fusions | Cohort B-ID: All Other FGF/FGFR Alterations | Other-ID | Cohort A-CD: FGFR3 Mutations or Fusions | Other-CD | Total
Number analyzed (Participants) | 103 | 44 | 9 | 101 | 3 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (9.09) | 65.1 (10.83) | 69.3 (7.98) | 68.5 (9.39) | 60.3 (9.02) | 67.5 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 14 | 1 | 23 | 1 | 68
  Male | 74 | 30 | 8 | 78 | 2 | 192
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 64 | 29 | 6 | 63 | 2 | 164
  Black or African-American | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 2 | 2 | 0 | 12 | 1 | 17
  Turkish | 1 | 0 | 0 | 0 | 0 | 1
  Persian | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 30 | 13 | 1 | 22 | 0 | 66
  Missing | 6 | 0 | 0 | 4 | 0 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 2 | 0 | 3
  Not Hispanic or Latino | 64 | 32 | 7 | 66 | 2 | 171
  Not Reported | 23 | 11 | 2 | 22 | 1 | 59
  Unknown | 5 | 1 | 0 | 3 | 0 | 9
  Captured as Other | 5 | 0 | 0 | 6 | 0 | 11
  Missing | 5 | 0 | 0 | 2 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in Participants With FGFR3 Mutations or Fusions on a CD Regimen
Description: ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) at any post-Baseline visit prior to first progressive disease (PD), per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1). CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. Response was based on review of scans by an independent centralized radiological review committee. Response was confirmed.
Time Frame: up to 1138 days
Population: Efficacy Evaluable Population: all participants enrolled in the study who had a known FGF/FGFR alteration confirmed by the sponsor's central laboratory and who had received at least 1 dose of study drug. The confidence interval was calculated based on the exact method for binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A-ID: FGFR3 Mutations or Fusions | Cohort B-ID: All Other FGF/FGFR Alterations | Other-ID | Cohort A-CD: FGFR3 Mutations or Fusions | Other-CD
Number analyzed (Participants) | 0 | 0 | 0 | 101 | 0
percentage of participants |  |  |  | 17.8 [10.92 to 26.70] |

2. Secondary Outcome: ORR in Participants With FGFR3 Mutations or Fusions on an ID Regimen
Description: ORR was defined as the percentage of participants with a best overall response of CR or PR at any post-Baseline visit prior to first PD, per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. Response was based on review of scans by an independent centralized radiological review committee. Response was confirmed.
Time Frame: up to 817 days
Population: Efficacy Evaluable Population. The confidence interval was calculated based on the exact method for binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A-ID: FGFR3 Mutations or Fusions | Cohort B-ID: All Other FGF/FGFR Alterations | Other-ID | Cohort A-CD: FGFR3 Mutations or Fusions | Other-CD
Number analyzed (Participants) | 103 | 0 | 0 | 0 | 0
percentage of participants | 23.3 [15.54 to 32.66] |  |  |  |

3. Secondary Outcome: ORR in Participants With All Other FGF/FGFR Alterations
Description: as for outcome 2
Time Frame: up to 1198 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A-ID: FGFR3 Mutations or Fusions | Cohort B-ID: All Other FGF/FGFR Alterations | Other-ID | Cohort A-CD: FGFR3 Mutations or Fusions | Other-CD
Number analyzed (Participants) | 0 | 44 | 0 | 0 | 0
percentage of participants |  | 6.8 [1.43 to 18.66] |  |  |

4. Secondary Outcome: ORR in All Participants on an ID or CD Regimen in Combined Cohorts
Description: as for outcome 2
Time Frame: up to 1198 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort A-ID + Cohort B-ID: Participants with FGFR3 mutations or fusions (Cohort A) or with all other FGF/FGFR alterations (Cohort B) self-administered oral pemigatinib at a starting dose of 13.5 mg QD on an ID (2-weeks-on/1-week-off therapy) schedule in 21-day cycles. Participants who did not reach the target serum phosphate level of > 5.5 mg/dL could have increased the daily dose to 18 mg, provided they had no ongoing Grade 2 or higher treatment-related TEAEs, and they had been compliant with taking the study drug.
- Cohort A-ID + Cohort A-CD: Participants with FGFR3 mutations or fusions self-administered oral pemigatinib at a starting dose of 13.5 mg QD on an ID (2-weeks-on/1-week-off therapy) schedule (Cohort A-ID) or on a CD (no planned dose hold) schedule (Cohort A-CD) in 21-day cycles. Participants who did not reach the target serum phosphate level of > 5.5 mg/dL could have increased the daily dose to 18 mg, provided they had no ongoing Grade 2 or higher treatment-related TEAEs, and they had been compliant with taking the study drug.
- Cohort A-ID + Cohort B-ID + Cohort A-CD: Participants with FGFR3 mutations or fusions (Cohort A) or with all other FGF/FGFR alterations (Cohort B) self-administered oral pemigatinib at a starting dose of 13.5 mg QD on an ID (2-weeks-on/1-week-off therapy) schedule (Cohort A-ID and Cohort B-ID) in 21-day cycles or on a CD (no planned dose hold) schedule (Cohort A-CD). Participants who did not reach the target serum phosphate level of > 5.5 mg/dL could have increased the daily dose to 18 mg, provided they had no ongoing Grade 2 or higher treatment-related TEAEs, and they had been compliant with taking the study drug.
Arm/Group | Cohort A-ID: FGFR3 Mutations or Fusions | Cohort B-ID: All Other FGF/FGFR Alterations | Other-ID | Cohort A-CD: FGFR3 Mutations or Fusions | Other-CD | Cohort A-ID + Cohort B-ID | Cohort A-ID + Cohort A-CD | Cohort A-ID + Cohort B-ID + Cohort A-CD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 147 | 204 | 248
percentage of participants |  |  |  |  |  | 18.4 [12.47 to 25.59] | 20.6 [15.26 to 26.79] | 18.1 [13.55 to 23.52]

5. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results occurring after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or required changes in the study drug(s). A TEAE was any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug and within 30 days of the last dose of study drug.
Time Frame: up to approximately 25 weeks
Population: Safety Population: all participants enrolled in the study who had received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A-ID: FGFR3 Mutations or Fusions | Cohort B-ID: All Other FGF/FGFR Alterations | Other-ID | Cohort A-CD: FGFR3 Mutations or Fusions | Other-CD
Number analyzed (Participants) | 103 | 44 | 9 | 101 | 3
Participants | 103 | 44 | 9 | 100 | 3

6. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the length of time from the start of the study drug (Day 1) to the earlier of death or disease progression by RECIST v1.1, as assessed by the independent centralized radiological review committee.
Time Frame: up to 1138 days
Population: Efficacy Evaluable Population. The "Other-ID" and "Other-CD" treatment groups were not included in the Efficacy Evaluable Population. The 95% confidence interval was calculated using the Brookmeyer and Crowley's method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A-ID: FGFR3 Mutations or Fusions | Cohort B-ID: All Other FGF/FGFR Alterations | Other-ID | Cohort A-CD: FGFR3 Mutations or Fusions | Other-CD
Number analyzed (Participants) | 103 | 44 | 0 | 101 | 0
months | 4.27 [3.91 to 6.05] | 2.04 [1.87 to 2.17] |  | 4.04 [3.45 to 4.17] |

7. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first overall response contributing to an objective response (CR or PR) to the earlier of death or first overall response of PD occurring after the first overall response contributing to the objective response. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. Response was based on review of scans by an independent centralized radiological review committee. Response was confirmed
Time Frame: up to 1075 days
Population: Efficacy Evaluable Population. The "Other-ID" and "Other-CD" treatment groups were not included in the Efficacy Evaluable Population. Only participants with a CR or PR were analyzed. The 95% confidence interval was calculated using the Brookmeyer and Crowley's method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A-ID: FGFR3 Mutations or Fusions | Cohort B-ID: All Other FGF/FGFR Alterations | Other-ID | Cohort A-CD: FGFR3 Mutations or Fusions | Other-CD
Number analyzed (Participants) | 24 | 3 | 0 | 18 | 0
months | 6.21 [4.60 to 7.95] | 10.02 [8.38 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. |  | 6.23 [4.14 to 8.25] |

8. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the length of time from the start of the study drug (Day 1) until the date of death due to any cause.
Time Frame: up to 1610 days
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A-ID: FGFR3 Mutations or Fusions | Cohort B-ID: All Other FGF/FGFR Alterations | Other-ID | Cohort A-CD: FGFR3 Mutations or Fusions | Other-CD
Number analyzed (Participants) | 103 | 44 | 0 | 101 | 0
months | 8.90 [7.46 to 15.18] | 9.13 [5.52 to 17.05] |  | 6.80 [5.26 to 9.10] |

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for up to approximately 25 weeks; All-cause Mortality was assessed for up to 1610 days.
Description: Treatment-emergent adverse events, defined as adverse events either reported for the first time or the worsening of pre-existing events after the first dose of study drug and within 30 days of the last dose of study drug, have been reported.
Arm/Group | Cohort A-ID: FGFR3 Mutations or Fusions | Cohort B-ID: All Other FGF/FGFR Alterations | Other-ID | Cohort A-CD: FGFR3 Mutations or Fusions | Other-CD
All-Cause Mortality (participants affected / at risk) | 88/103 | 39/44 | 8/9 | 83/101 | 2/3
Serious Adverse Events (participants affected / at risk) | 45/103 | 26/44 | 3/9 | 48/101 | 1/3
Other Adverse Events (participants affected / at risk) | 101/103 | 43/44 | 9/9 | 99/101 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A-ID: FGFR3 Mutations or Fusions (N=103) | Cohort B-ID: All Other FGF/FGFR Alterations (N=44) | Other-ID (N=9) | Cohort A-CD: FGFR3 Mutations or Fusions (N=101) | Other-CD (N=3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chorioretinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Detachment of retinal pigment epithelium (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder enlargement (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 5 (5) | 3 (3) | 0 (0) | 5 (5) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Optic neuropathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral nerve paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyp (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomal hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (6) | 1 (1) | 0 (0) | 8 (11) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urostomy complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasculitis necrotising (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral oesophagitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A-ID: FGFR3 Mutations or Fusions (N=103) | Cohort B-ID: All Other FGF/FGFR Alterations (N=44) | Other-ID (N=9) | Cohort A-CD: FGFR3 Mutations or Fusions (N=101) | Other-CD (N=3)
Abdominal pain (Gastrointestinal disorders) | 20 (28) | 11 (12) | 1 (1) | 7 (9) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 3 (4) | 0 (0) | 6 (7) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 5 (6) | 1 (1) | 4 (4) | 0 (0)
Ageusia (Nervous system disorders) | 6 (6) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 9 (11) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 49 (50) | 16 (16) | 7 (7) | 38 (38) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 19 (22) | 10 (10) | 1 (1) | 18 (19) | 0 (0)
Anxiety (Psychiatric disorders) | 5 (6) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arcus lipoides (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (22) | 6 (7) | 1 (1) | 19 (22) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (6) | 0 (0) | 0 (0) | 7 (8) | 0 (0)
Asthenia (General disorders) | 28 (31) | 9 (9) | 2 (2) | 32 (37) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (22) | 6 (6) | 2 (2) | 15 (15) | 1 (1)
Blepharitis (Eye disorders) | 8 (10) | 1 (1) | 0 (0) | 9 (9) | 1 (1)
Blood creatinine increased (Investigations) | 17 (19) | 5 (5) | 2 (2) | 20 (22) | 1 (1)
Blood phosphorus increased (Investigations) | 9 (11) | 4 (6) | 2 (2) | 13 (23) | 1 (1)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 6 (7) | 1 (1) | 0 (0) | 6 (6) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 4 (5) | 2 (2) | 1 (1) | 6 (6) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 36 (46) | 11 (13) | 4 (4) | 33 (35) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Corneal neovascularisation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 3 (3) | 0 (0) | 5 (5) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 32 (38) | 11 (12) | 4 (4) | 29 (33) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 8 (12) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Detachment of macular retinal pigment epithelium (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 53 (89) | 19 (28) | 6 (8) | 34 (55) | 2 (2)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 12 (14) | 4 (4) | 1 (2) | 4 (6) | 0 (0)
Dry eye (Eye disorders) | 21 (27) | 7 (7) | 4 (4) | 19 (20) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 33 (35) | 13 (13) | 7 (7) | 39 (39) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 21 (23) | 6 (6) | 4 (5) | 22 (23) | 2 (2)
Dysgeusia (Nervous system disorders) | 32 (35) | 9 (10) | 6 (6) | 31 (33) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 10 (16) | 1 (1) | 2 (2) | 7 (7) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 4 (5) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (6) | 1 (1) | 4 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4) | 1 (1) | 5 (5) | 1 (1)
Dysuria (Renal and urinary disorders) | 4 (5) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 3 (3) | 2 (2) | 14 (18) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye haematoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Eyelid pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 36 (44) | 16 (17) | 3 (3) | 29 (33) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 7 (7) | 0 (0)
Gingivitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 8 (11) | 6 (7) | 2 (2) | 12 (15) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 5 (5) | 0 (0) | 5 (5) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 11 (12) | 1 (2) | 1 (1) | 7 (8) | 0 (0)
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (7) | 4 (7) | 0 (0) | 8 (11) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 35 (39) | 13 (15) | 4 (4) | 56 (95) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (8) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (9) | 6 (10) | 1 (1) | 9 (12) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 13 (20) | 3 (4) | 1 (2) | 4 (4) | 0 (0)
Hypotension (Vascular disorders) | 10 (11) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypouricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 2 (2) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 12 (13) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 4 (4) | 1 (1) | 2 (2) | 5 (5) | 0 (0)
Lacrimation increased (Eye disorders) | 2 (3) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (3) | 6 (7) | 0 (0) | 1 (1) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Meibomian gland dysfunction (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 1 (1) | 5 (5) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 (11) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5) | 1 (1) | 10 (10) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 8 (9) | 2 (2) | 0 (0) | 10 (11) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 7 (8) | 2 (2) | 1 (1) | 6 (6) | 0 (0)
Nail toxicity (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1) | 0 (0) | 7 (7) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 28 (39) | 13 (17) | 1 (1) | 18 (19) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 6 (6) | 8 (9) | 0 (0) | 10 (10) | 0 (0)
Onychalgia (Skin and subcutaneous tissue disorders) | 4 (6) | 2 (2) | 0 (0) | 6 (6) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 10 (10) | 6 (7) | 0 (0) | 10 (10) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 6 (7) | 3 (3) | 1 (1) | 8 (8) | 0 (0)
Oral candidiasis (Infections and infestations) | 3 (4) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 5 (5) | 4 (5) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3) | 0 (0) | 5 (5) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 6 (6) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (14) | 4 (5) | 1 (1) | 15 (18) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 (10) | 3 (3) | 1 (1) | 28 (31) | 0 (0)
Paronychia (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 8 (10) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Proteinuria (Renal and urinary disorders) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Punctate keratitis (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 7 (8) | 0 (0)
Pyrexia (General disorders) | 14 (19) | 6 (6) | 0 (0) | 12 (17) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2) | 0 (0) | 8 (8) | 0 (0)
Retinal detachment (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 9 (9) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 48 (70) | 13 (14) | 3 (3) | 45 (56) | 1 (1)
Subretinal fluid (Eye disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trichiasis (Eye disorders) | 6 (6) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Trichomegaly (Eye disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 25 (31) | 10 (16) | 1 (1) | 10 (12) | 0 (0)
Vision blurred (Eye disorders) | 6 (7) | 1 (3) | 1 (1) | 7 (8) | 0 (0)
Visual acuity reduced (Eye disorders) | 5 (5) | 0 (0) | 0 (0) | 10 (10) | 0 (0)
Visual impairment (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Vitamin D decreased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 4 (5) | 1 (1) | 1 (1) | 2 (2) | 1 (2)
Vomiting (Gastrointestinal disorders) | 19 (29) | 10 (15) | 0 (0) | 12 (19) | 1 (1)
Weight decreased (Investigations) | 19 (21) | 2 (2) | 1 (1) | 12 (12) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/14/NCT02872714/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT02872714/SAP_001.pdf